CLINICAL TRIAL: NCT00612534
Title: A Multicenter, Randomized, Placebo-Controlled Phase 2 Study to Evaluate the Clinical Efficacy, Safety, and Tolerability of ARX-F01 Sublingual Sufentanil in Patients Undergoing Elective Unilateral Total Knee Replacement
Acronym: ARX-F01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARX-C-001
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Sufentanil NanoTab
- 2 (Experimental)
  Interventions: Drug: Sufentanil NanoTab
- 3 (Experimental)
  Interventions: Drug: Sufentanil NanoTab
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo NanoTab

INTERVENTIONS:
Drug: Sufentanil NanoTab — 5 mcg Sufentanil NanoTab taken sublingually q 20 minutes as needed for pain for 12 hours
  Other Names: ARX-F01
  Arms: 1
Drug: Placebo NanoTab — Placebo NanoTab taken sublingually q 20 minutes as needed for pain for 12 hours
  Arms: 4
Drug: Sufentanil NanoTab — 10 mcg Sufentanil NanoTab taken sublingually q 20 minutes as needed for pain for 12 hours
  Other Names: ARX-F01
  Arms: 2
Drug: Sufentanil NanoTab — 15 mcg Sufentanil NanoTab taken sublingually q 20 minutes as needed for pain for 12 hours
  Other Names: ARX-F01
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate three different dosage strengths of sublingual ARX-F01 (Sufentanil NanoTab) versus a sublingual Placebo NanoTab for the treatment of post-operative pain in subjects following total knee replacement surgery. We hypothesize that subjects receiving placebo will have poor pain relief and will drop out of the study sooner and more often than the ARX-F01-treated subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 45 to 80 years of age.
* Patient is scheduled for an elective, unilateral, unicondylar, bi- or tri-compartmental, cemented or uncemented knee replacement under general or spinal anesthesia that does not include use of an intrathecal opioid.
* Patient must be classified as American Society of Anesthesiologists (ASA) class I - III.
* Patient must have Body Mass Index [BMI = weight (kg)/height (m2)] between 18 and 39, inclusively.
* Female patients of childbearing potential must be using an effective method of birth control from the screening visit through the end of study. Acceptable methods of birth control include oral or transdermal contraceptives, condom, spermicidal foam, intrauterine device (IUD), progestin implant or injection, abstinence, vaginal ring, or sterilization of partner. The reason for non-childbearing potential, such as bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or postmenopausal for ≥1 year, must be specified in the patient's case report form (CRF).
* The patient must be willing and able to understand the study procedures and the use of pain scales, and to communicate meaningfully with the study personnel.
* The patient must provide written informed consent and sign the Informed Consent approved by the Institutional Review Board (IRB).

Exclusion Criteria:

* Patient has previously undergone a knee replacement of the same knee.
* A passive range-of-motion (PRM) will be used before the 12-hour study period is complete
* Patient has previously not responded to opioid analgesics for treatment of pain.
* Patient is currently taking or has taken an opioid for more than 30 consecutive days of daily use at a daily dose equivalent to greater than 15 mg morphine within the past 3 months prior to surgery (e.g. more than 3 doses per day of Vicodin®, Norco®, Lortab® with 5 mg hydrocodone per tablet).
* Patient has an allergy or hypersensitivity to opioids.
* Patient currently has sleep apnea that has been documented by a sleep laboratory study.
* Patient has any screening laboratory test value outside the laboratory normal range which is considered clinically significant by the Investigator.
* Patient has a contraindication to the use of general anesthesia.
* Patient is a woman who is pregnant or lactating.
* Patient has psychiatric disease or encephalopathy severe enough to prevent patient from providing reliable study documentation.
* Patient, in the Investigator's judgment, does not have adequate ability to read and understand English.
* Patient has a medical condition that, in the Investigator's opinion, could adversely impact the patient's participation or safety, conduct of the study, or interfere with the pain assessments, including fracture or active infection.
* Patient has clinically significant renal or liver impairment which could affect metabolism or clearance of sufentanil.
* Patient has a painful physical condition other than knee arthritis that, in the opinion of the Investigator, may confound post-operative pain assessments.
* Patient has a history of drug, prescription medicine, or alcohol abuse within the past 2 years or a positive test for drugs of abuse at screening.
* Patient is receiving oxygen therapy at the time of screening.
* Patient participated in a clinical trial of an investigational drug or device within 30 days of screening visit or is scheduled to receive an investigational product other than ARX-F01 while participating in this study.

Exclusion Criteria at Randomization (during early PACU time period):

* Patient has a respiratory rate that is less than 8 breaths per minute or greater than 24 breaths per minute,
* Patient has arterial oxygen saturation by pulse oximetry (SpO2) of less than 90% with supplemental oxygen.
* Patient is not able to answer questions and follow commands.
* Patient has vomiting that is not responsive to standard treatment.
* The surgical procedure from incision to closure was longer than 3 hours.
* There have been any deviations from the surgical or anesthetic protocols as specified in the protocol.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Trio Clinical Research, Durham, North Carolina, United States

REFERENCES:
- [Result] Minkowitz HS, Singla NK, Evashenk MA, Hwang SS, Chiang YK, Hamel LG, Palmer PP. Pharmacokinetics of sublingual sufentanil tablets and efficacy and safety in the management of postoperative pain. Reg Anesth Pain Med. 2013 Mar-Apr;38(2):131-9. doi: 10.1097/AAP.0b013e3182791157. PMID 23271030

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sufentanil NanoTab 5 Mcg | Sufentanil NanoTab 10 Mcg | Sufentanil NanoTab 15 Mcg | Placebo NanoTab
Started | 24 | 26 | 20 | 24
Completed | 11 | 9 | 13 | 7
Not Completed | 13 | 17 | 7 | 17
Not completed — Adverse Event | 0 | 4 | 2 | 1
Not completed — Lack of Efficacy | 13 | 12 | 5 | 16
Not completed — Other Reason | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sufentanil NanoTab 5 Mcg | Sufentanil NanoTab 10 Mcg | Sufentanil NanoTab 15 Mcg | Placebo NanoTab | Total
Number analyzed (Participants) | 24 | 26 | 20 | 24 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.0) | 64.6 (9.6) | 62.5 (8.0) | 63.3 (7.6) | 62.8 (8.7)
Age, Customized [Number; unit: participants]
  <40 years | 0 | 0 | 0 | 0 | 0
  40 to 64 years | 15 | 12 | 10 | 11 | 48
  >=65 years | 9 | 14 | 10 | 13 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 12 | 11 | 50
  Male | 9 | 14 | 8 | 13 | 44
Region of Enrollment [Number; unit: participants]
  United States | 24 | 26 | 20 | 24 | 94

OUTCOME MEASURES:

1. Primary Outcome: SPID-12
Description: SPID-12 is the sum of the pain intensity difference (PID) over the 12 hour time period. A pain intensity score of 0 (no pain) to 10 (worst possible pain) is obtained before starting the study and throughout the 12 hour time period. The pain score at each assessment time point is subtracted from the baseline pain score (starting point) to provide the total sum score or SPID-12. A higher SPID-12 score is better and indicates a reduction in pain intensity compared to the baseline score. Per protocol, pain scores are collected at 15 different time points. If all scores are collected, the full range of SPID-12 scores could be -150 to 150.
Time Frame: 12 hours after first dose
Population: One patient in Sufentanil NanoTab 10 mcg group received the incorrect treatment so was not included in efficacy analysis
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sufentanil NanoTab 5 Mcg | Sufentanil NanoTab 10 Mcg | Sufentanil NanoTab 15 Mcg | Placebo NanoTab
Number analyzed (Participants) | 24 | 25 | 20 | 24
units on a scale | 2.87 (5.68) | 1.28 (5.60) | 12.66 (6.25) | -7.39 (5.71)
Statistical Analysis 1: Comparison: Sufentanil NanoTab 5 Mcg vs Placebo NanoTab; Test type: Superiority or Other; p = 0.194, ANCOVA; Mean Difference (Final Values) = 10.26, 95% CI [-5.32 to 25.83], Standard Error of Mean 7.83
Statistical Analysis 2: Comparison: Sufentanil NanoTab 10 Mcg vs Placebo NanoTab; Test type: Superiority or Other; p = 0.268, ANCOVA; Mean Difference (Final Values) = 8.67, 95% CI 2-sided [-6.78 to 24.11], Standard Error of Mean 7.77
Statistical Analysis 3: Comparison: Sufentanil NanoTab 15 Mcg vs Placebo NanoTab; Test type: Superiority or Other; p = 0.018, ANCOVA; Mean Difference (Final Values) = 20.05, 95% CI 2-sided [3.54 to 36.56], Standard Error of Mean 8.30

ADVERSE EVENTS:
Arm/Group | Sufentanil NanoTab 5 Mcg | Sufentanil NanoTab 10 Mcg | Sufentanil NanoTab 15 Mcg | Placebo NanoTab
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/26 | 1/20 | 1/24
Other Adverse Events (participants affected / at risk) | 13/24 | 12/26 | 10/20 | 8/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sufentanil NanoTab 5 Mcg (N=24) | Sufentanil NanoTab 10 Mcg (N=26) | Sufentanil NanoTab 15 Mcg (N=20) | Placebo NanoTab (N=24)
acute renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — not related to study drug
chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — not related to study drug
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — not related to study drug
hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — not related to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sufentanil NanoTab 5 Mcg (N=24) | Sufentanil NanoTab 10 Mcg (N=26) | Sufentanil NanoTab 15 Mcg (N=20) | Placebo NanoTab (N=24)
nausea (Gastrointestinal disorders) | 7 | 9 | 4 | 5
vomiting (Gastrointestinal disorders) | 2 | 4 | 3 | 1
somnolence (Nervous system disorders) | 1 | 0 | 2 | 1
respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
neutrophil count increased (Investigations) | 1 | 0 | 0 | 1
dizziness (Nervous system disorders) | 3 | 1 | 1 | 0
white blood cell count increased (Investigations) | 1 | 0 | 0 | 1
hypotension (Vascular disorders) | 0 | 1 | 0 | 1
bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 — All adverse events in this table were assessed by the PI as possibly or probably related to study drug
tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
fatigue (General disorders) | 0 | 0 | 0 | 1
pyrexia (General disorders) | 0 | 0 | 0 | 1
lymphocyte count increased (Investigations) | 0 | 0 | 0 | 1
pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
oxygen saturation decreased (Investigations) | 0 | 1 | 1 | 0
headache (Nervous system disorders) | 0 | 0 | 2 | 0
oral mucosal discoloration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 0 | 0
lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
prior written consent of sponsor